CLINICAL TRIAL: NCT04315584
Title: FDG and FDOPA PET Demonstration of Functional Brain Abnormalities
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Bijoy Kundu, Bijoy Kundu, PhD, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSR190096
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Glioblastoma
Keywords: glioblastoma; PET; CT; multiparametric MRI; brain imaging; tumor recurrence
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; fluorodopa F 18

STUDY DESIGN:
Intervention Model Description: All 5 study subjects will undergo the same procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Experimental): Study subjects will receive 18FDG via an IV before undergoing one PET/CT scan over 60 minutes. They will then receive an IV injection of Gadovist for contrast before undergoing a multiparametric MRI scan. Subjects will also receive (18)F-FDOPA via an IV before undergoing another PET/CT scan over 60 minutes.
  Interventions: Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Multiparametric Magnetic Resonance Imaging Scan; Radiation: Fludeoxyglucose F-18; Radiation: fluorine F 18 fluorodopa

INTERVENTIONS:
Procedure: Positron Emission Tomography — Undergo PET/CT Scans
  Other Names: PET; PET Scan; Positron Emission Tomography Scan; Medical Imaging, Positron Emission Tomography
Procedure: Computed Tomography — Undergo PET/CT Scans
  Other Names: CT; CT Scan; Computerized Axial Tomography; CAT; CAT scan
Procedure: Multiparametric Magnetic Resonance Imaging Scan — Undergo a multiparametric MRI scan
  Other Names: mpMRI; multiparametric MRI
Radiation: Fludeoxyglucose F-18 — IV (intravenous) administration of radiotracer
  Other Names: FDG; 18 FDG; fludeoxyglucose F 18; 2-F18-fluoro-2-deoxy-D-glucose; 2-F18-fluoro-2-deoxyglucose
Radiation: fluorine F 18 fluorodopa — IV (intravenous) administration of radiotracer
  Other Names: 18F-6- L-fluorodopa; 18F-DOPA; 18F-FDOPA; 3,4-dihydroxy-6-(18)F-fluoro-l-phenylalanine; L-6-[ 18F]fluoro-3, 4-dihydroxyphenylalanine; (18)F-FDOPA

SUMMARY:
The purpose of this pilot study will be to conduct a clinical trial using a time-of-flight PET scanner and MRI scanner to test an improved method for differentiating tumor recurrence from radiation necrosis in glioblastoma patients. We will attempt to do so by performing a static and dynamic FDG-PET scan, a static and dynamic FDOPA-PET scan, and a multiparametric MRI scan - then comparing the results with surgical pathology and static FDG-PET scans. We hypothesize that the new quantitative kinetic analytical methods using FDOPA in combination with FDG will provide crucial functional information to distinguish recurrent tumors from treatment-induced radiation changes in patients with treated brain neoplasms. This is important for improving patient outcomes by allowing treating physicians to more accurately tailor treatments. Furthermore, dynamic FDG and FDOPA PET will be combined with high resolution anatomic and physiologic MRI in order to develop a multimodal multiparametric approach for differentiating tumor recurrence from treatment effect.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective will be to evaluate the diagnostic accuracy of Dynamic PET imaging in differentiating tumor recurrence from treatment effect (radiation necrosis or pseudoprogression) in patients previously treated with chemo-radiation therapy for primary high grade gliomas. This will be accomplished by examining the concordance between the Dynamic PET imaging prediction and the criterion standard, which will be based on either surgical pathology or an integrated clinical/MRI determination within a 3-6 month interval after Dynamic PET imaging.

SECONDARY OBJECTIVES:

I. The diagnostic accuracy of Static PET imaging, advanced MRI, and advanced MRI + Dynamic PET imaging in differentiating tumor recurrence from radiation-induced necrosis in high grade glioma patients will be examined in the same exact way as just outlined for Dynamic PET imaging.

OUTLINE:

Subjects receive 18FDG (first scan) and (18)F-FDOPA (2-14 days from the first scan) intravenously (IV) slowly over a period of 15-20 seconds and then undergo dynamic PET scans over a period of 60-90 minutes. CT scans on the subjects are performed before the dynamic PET scans for 5 minutes. Subjects also undergo MRI brain examinations just prior to the FDOPA scan over a period of 1 hour, which includes T1 weighed, T1 weighted contrast enhanced, T2 weighted, Diffusion tensor imaging, MR spectroscopy, and Dynamic susceptibility contrast perfusion weighted (DSC-PWI) imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Known or suspected recurrent malignant brain tumors
* Radiographic worsening reported on MRI shortly (within 3 months) after completion of radiation and temozolomide therapy
* Able to lie flat and/or still for a minimum of 60 minutes
* Willingness and ability to comply with scheduled visits and study procedures
* Patients who have a clinical indication for a PET-CT
* If female, patient must be postmenopausal or surgically sterile

Exclusion Criteria:

- Conditions that preclude a clinical brain FDG PET study, including: Consumption of liquids with sugar and/or caffeine prior to the study, Blood glucose levels over 150 mg/mL, Eating or drinking calories of any type within 4 hours of radiotracer injection, Hyperinsulinemia, Patients who for any reason cannot tolerate lying supine for 60 minutes

* Conditions that preclude a FDOPA PET study, including: Consuming a diet that is NOT low in protein after the previous evening meal
* Tumor located in the striatum
* Changes in medication (new prescriptions or change in dosages) between visits 1 and 2
* Pregnant, nursing, or lactating
* Women of childbearing potential (premenopausal female capable of becoming pregnant), which also includes:

women on oral, injectable, or mechanical contraceptives, women who are single, women whose male partners have been vasectomized or whose male partners have received or are utilizing mechanical contraceptive devices

* Weight > 450 lbs
* Known allergic reactions to 3,4-dihydroxy-6-[18F]fluoro-L-phenylalanine (18F-FDOPA) and Fluorine-18 fluorodeoxyglucose (18F-FDG)
* Confirmation that study eligibility criteria have not been met between visits 1 and 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Quantitative parametric maps indicating differences in rates of glucose and amino acid uptake (Ki) obtained from dynamic FDG and FDOPA scans respectively. | Up to 6 months
  Will be derived from PET/CT scan imaging.
Quantitative parametric maps indicating differences in details (d) components of the wavelet transform analysis, d6 and d8, based on established tumor feature criterions. | Up to 6 months
  Will be derived from MRI brain scan imaging.
Semi-quantitative standardize uptake value (SUV) parametric maps based on static PET scans (last 20 minutes of the dynamic PET scans). | Up to 6 months
  Will be derived from PET/CT scan imaging.
MRI brain metrics | Up to 6 months
  Including anatomic assessment based on T1, T2, and contrast enhanced T1 weighted imaging, MR spectroscopy data (choline, creatinine, and N-acetyl acetate peak integrals and ratios), MR perfusion data (relative cerebral blood volume), and diffusion tensor imaging data (apparent diffusion coefficient, fractional anisotropy)
Surgical pathology or 3-6 month interval multidisciplinary clinical evaluation. | Up to 6 months
  To be compared with the imaging analyses for comparing ability to differentiate tumor recurrence from radiation necrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Bijoy Kundu, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No